CLINICAL TRIAL: NCT01954914
Title: Plerixafor as a Salvage Regimen to Mobilize Allogeneic Stem Cells in Healthy Volunteers
Acronym: MOBIL1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: University Hospital Carl Gustav Carus (Other); Cellex Gesellschaft für Zellgewinnung mbH Dresden (Unknown); Cellex Gesellschaft für Zellgewinnung mbH Köln (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-MOBIL1-056
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Blood Stem Cell Harvest Failure
Keywords: Plerixafor; donor; allogeneic peripheral stam cell donation; PBSC; poor donors
MeSH Terms: interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plerixafor, Mozobil (Experimental): Administration of a single dose of Plerixafor 240 µg/kg body weight of the donor SC in the evening at 10 PM after frustraneous stem cell apheresis on day 1.
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Administration of a single dose of Plerixafor 240 µg/kg body weight of the donor SC in the evening at 10 PM after frustraneous stem cell apheresis on day 1.
  Other Names: Mozobil

SUMMARY:
With a standard mobilization regimen using G-CSF, approximately 5% of allogeneic donors does not mobilize enough CD34+ cells to reach an optimal dose for transplantation and are therefore called "poor mobilizers". A generally accepted optimum CD34+ PBSC dose for allogeneic transplantation is > 4.5 x 106/kg body weight of the recipient. The minimum total CD34+ PBSC dose certainly amounts to 2 x 106/kg body weight of the recipient.The objective of this trial is to assess the efficacy of a single dose of Plerixafor as salvage procedure in allogeneic stem cell donors with a poor CD34+ cell yield after the first day of peripheral blood stem cell collection.

DETAILED DESCRIPTION:
In this trial the administration of a single dose of Plerixafor 240 µg/kg body weight of the donor SC in the evening at 10 PM after frustraneous stem cell apheresis on day 1 will be provided. The apheresis on day 2 is performed according to standard recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Donor age between 18 years and 75 years
* Eligibility of the donor for allogeneic PBSC donation according to German Guidelines (Richtlinien Hämotherapie Bundesärztekammer 2005) preceding the application of G-CSF
* The donor has understood and signed the donor information. Written informed consent has been obtained.
* Donation of less than 2.0 x 106 CD34 cells/kg recipient body weight after one apheresis following five days of stem-cell mobilization with Lenograstim 7.5 to 10 µg/kg donor body weight
* First leukapheresis according to standard recommendations with a processing of 3 x donor's blood volume ± 10% using either of the following three devices: Cobe Spectra (Terumo BCT) Spectra Optia (Terumo BCT) Fresenius COM.TEC

Exclusion Criteria:

* Pain or any discomfort in the left upper square of the abdomen during physical examination immediately prior to study inclusion or any spontaneous complaint about abdominal discomfort without an ultrasound investigation which rules out splenomegaly.
* Palpitations or any thoracic discomfort in the absence of an ECG which shows normal results
* Platelet count < 80 x 109/l
* Serum creatinine > 80 µmol/l for female donors or > 106 µmol/l for male donors. If serum creatinine is elevated then the estimated creatinine clearance has to be > 50 ml/min. Estimation by the Modification of Diet in Renal Disease equation where predicted GFR(ml/min/1.73m2) = 186 x (Serum Creatinine in mg/dL)-1.154 x (age in years)-0.203 x (0.742 if patient is female) x (1.212 if patient is black) or GFR(ml/min/1.73m2) = 186 x 176 (Serum Creatinine in µmol/l)-1.154 x (age in years)-0.203 x (0.742 if patient is female) x (1.212 if patient is black)
* Contraindications against a second leukapheresis, such as severe side effects during 1st leukapheresis (intolerable pain, severe circulatory disorder, severe citrate intolerance)
* Missing written approval by the transplant center that the transplantation of the Plerixafor-mobilized graft is being considered
* Treatment with any known non-marketed drug substance or experimental therapy within 4 weeks prior to enrolment or participation in any other interventional clinical study
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise donor safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Female donors of childbearing potential unable or unwilling to use adequate contraception methods for three months after the administration of the study drug. Adequate methods for contraception in female donors are sexual abstinence, the use of condoms by their partners, vasectomy of the partner or hormonal contraception.
* Male donors unable or unwilling to use adequate contraception methods for one month after the administration of the study drug. Adequate methods for contraception for males are sexual abstinence or the use of condoms.
* Known intolerance to Plerixafor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Rate of donation success | 1 day
  A generally accepted optimum CD34+ PBSC dose for allogeneic transplantation is > 4.5 x 10e6/kg body weight of the recipient. The minimum total CD34+ PBSC dose certainly amounts to 2 x 10e6/kg body weight of the recipient.

SECONDARY OUTCOMES:
Assessment of donor safety and tolerability based on self-reporting on a questionnaire, clinical findings, and laboratory evaluations; and evaluation of the cellular composition of the apheresis products collected with and without Plerixafor application. | 30 days
  The composition of apheresis products collected after filgrastim or filgrastim plus Plerixafor will be characterized with respect to:
  * CD34+ cell subsets (differential expression of prominin1/CD133+)33
  * Regulatory T-cells34
  * Dendritic cells
  * Myeloid-derived suppressor cells

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Hölig, Dr. med., Principal Investigator — Universitätsklinikum Carl Gustav Carus, Medizinische Klinik und Poliklinik I, 01307 Dresden
Locations (3):
- Germany (3):
  - Cellex Gesellschaft für Zellgewinnung mbH Köln, Cologne
  - Cellex Gesellschaft für Zellgewinnung mbH Dresden, Dresden
  - Universitätsklinikum Dresden, Medizinische Klinik I, Dresden

IPD SHARING:
Plan to Share IPD: No